CLINICAL TRIAL: NCT04921410
Title: Artificially Intelligent Biofeedback Sleeve for Prevention and Rehabilitation of Traumatic Knee Injury
Brief Title: AI Driven Biofeedback Wearable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Clifton R. Haider, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-004218
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Knee Injuries
Keywords: injury; prevention; biofeedback; knee; wearable; rehabilitation
MeSH Terms: conditions — Knee Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Sleeve Effects on Preventive Biomechanics (Experimental): Biofeedback wearable sleeve will be utilized in at least 2 groups of athletes. This randomized group will receive an 'active' wearable device. The device will be worn during regular sport practice sessions for 8-16 weeks. The device will provide haptic feedback directly associated with potentially injurious events as determined by previously established cut-off values and artificially-intelligent algorithms.
  Interventions: Device: Biofeedback Knee Sleeve
- Sham Biofeedback (Sham Comparator): Biofeedback wearable sleeve will be utilized in at least 2 groups of athletes. This randomized group will receive a 'sham' wearable device. The device will be worn during regular sport practice sessions for 8-16 weeks. The device will provide random feedback at random intervals not directly associated with potentially injurious events.
  Interventions: Device: Sham Biofeedback

INTERVENTIONS:
Device: Biofeedback Knee Sleeve — The biofeedback knee sleeve is a device that is artificially-intelligent and utilizes determined cut-off values of knee motion and forces to determine whether a motion is 'good' or 'bad'. A 'bad' knee motion will provide a haptic output to the wearer (biofeedback) so that they can take note of what the previous motion was that caused the device to signal a warning.
  Arms: Biofeedback Sleeve Effects on Preventive Biomechanics
Device: Sham Biofeedback — The biofeedback knee sleeve is a device that is artificially-intelligent and utilizes determined cut-off values of knee motion and forces to determine whether a motion is 'good' or 'bad'. This intervention will provide sham biofeedback during training sessions.
  Arms: Sham Biofeedback

SUMMARY:
The purpose of this study is to conduct a comprehensive clinical and biomechanical screening of high school, collegiate-level, recreational, and Olympic/professional-level athletes with the goal of identifying individual functional and performance deficits that lead to future injury.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 12 - 65 years old.
* Athlete at High School, Collegiate, Recreational, Olympic / Professional level.

Exclusion Criteria:

* Indidividual under 12 or over 65 years old.
* Lower extremity injury in the past 6 months.
* History of neurological disease, vestibular or visual disturbance.
* Any other pathology that would impair motor performance.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
3D Motion | 8-16 weeks
  Lower limb kinetics and kinematics will be calculated with inverse dynamics from 3D motion capture.
Rate / Incidence of Knee Injury | 8-16 weeks
  Knee injuries will be reported via coach, athletic trainer, or medical staff

SECONDARY OUTCOMES:
Landing force | 8-16 weeks
  Non-contact injuries to the lower limb are dependent on ground reaction force. As ground reaction force is minimized during landing, so is the risk for injury as lower forces are transmitted through the limb.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Haider, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials